# A PROSPECTIVE CONTROLLED MULTI-CENTER STUDY ON VANGUARD™ COMPLETE KNEE & VANGUARD™ HIGH FLEX RP KNEE

## **GENERAL INFORMATION**

## **Principal Investigators**

Yong In, M.D., Ph.D. – 75 Cases Chul-Won Ha, M.D., Ph.D. – 75 Cases Myung Chul Lee, M.D., Ph.D. – 75 Cases Seong-II Bin, M.D., Ph.D. – 75 Cases

Principal investigators are responsible for the overall project and performing the surgical procedures in all study groups. Responsible for applying for ethical and management approval, recruitment of patients, obtaining patient consent, managing postoperative care of patients and adverse event reporting.

## **Study Sponsor**

**Biomet Korea** 

Study sponsors take responsibility for initiation, management, and/or financing of a clinical studies at investigational sites.

## **Study Monitor in Korea**

Anna Lee

Study monitors are responsible for carrying out the monitoring procedure as indicated in the protocol.

## STUDY OBJECTIVE

The primary objectives of this clinical study include:

- Evaluate size fit and long term performance of Vanguard Complete Knee ("Fixed") System in Asian and Latino population Compare Vanguard High Flex Rotating Platform ("High Flex") Knee System to Vanguard Complete Knee System in Asian population in terms of:
  - Early ROM
  - Clinical outcomes
- Compare current design to new design of Vanguard High Flex Rotating Platform Knee System in terms of :
  - Early ROM
  - Clinical outcomes

#### **DEVICE DESCRIPTION**

## **Vanguard Complete Knee**

Vanguard Knee is a metal and polyethylene system designed to replace the body's natural knee joint and is indicated for cemented tibial and cementless femoral use. The system contains three (3) primary components and one (1) peripheral component. The primary components include, femoral, tibial, and bearing components, while the peripheral component is the patella button. The use of the patella button is optional.

# Vanguard High Flex Rotating Platform Knee (current design)

Vanguard High Flex RP knee is an extension to the existing Vanguard Knee and has been specifically designed to facilitate greater than 135 degrees of knee flexion as required by certain patients. Specifically the Vanguard High-Flex Knee components are required to be able to flex to 150° without point loading or falling off the back of the tibia and to be hyper extended to 15°. It should be noted that this range of motion would only be obtained where the patient had similar flexion and hyperextension ability prior to the arthroplasty. The decision on which rotating platform variant to use is at the discretion of the operating surgeon

Mobile bearing knees are considered advantages as they enable improved congruency between the femoral component and the bearing, compared with a fixed bearing, which results in lower contact stresses of the bearing, thereby reducing wear. Another advantage of mobile bearings is the ability for self-alignment, which reduces wear caused by mal-lalignment, enabling the knee to function more naturally and prevents torsion stress on the implant/bone cement/bone interface which may cause loosening.

The tibial tray of the High Flex knee is available in 9 sizes, from 59 to 91mm in 4 mm increments, in interkok finish for cemented applications or with porous plasma sprayed titanium coating for cementless use. It is manufactured from cast cobalt chromium alloy. The stem has a tapered cone geometry for press fit stability. In the cementless option the proximal 1/3 of the stem is porous coated with plasma sprayed titanium. (Note: The tibial trays are manufactured and CE marked by Biomet Spain).

The femoral component is offered in thirteen sizes from 55 to 80mm in 2.5 mm increment, it is anatomic in design (i.e. right and left). It is manufactured from cast cobalt chromium alloy.

The bearing is compression moulded UHMPWE (ArCom). It is matched to the femoral component and is available in 5 thickness from 10-18mm (2mm increments) and 13 sizes from 50mm to 80mm (2.5mm increments). The bearing was designed specifically for the High-Flex to allow rotation of ±8° without overhang.

The patella has an anatomic design and is matched to the thirteen sizes of femoral component patella tracks. It is available in of one thickness only. It is compression moulded from UHMWPE (ArCom). Use of the patella button is optional at the discretion of the surgeon.

05<sup>th</sup>-Nov-2014 2

# STUDY DESIGN

The study is designed as a prospective, controlled multi-center study including sites from Korea, Japan and Mexico.

To achieve all the primary objectives, the study will include 2 subgroups. The relationship between the two subgroups is illustrated in the following table and graph:

| Subgroup | Objectives | Trial<br>Group | Control Group | Design | Endpoint(s) |
|---|---|---|---|---|---|
| 2 | Compare early ROM, Clinical Outcomes, assess Kinetic and Kinematic characteristics between Vanguard Complete Knee System and Vanguard High Flex Rotating Platform Knee System* | Vanguard<br>Complete<br>Knee<br>System w/<br>std tray<br>(part of<br>subgroup<br>1 control) | Vanguard<br>High Flex RP<br>(Current<br>Design) | RCT | ROM, AKS,. |
| 4** | Compare early ROM, clinical outcomes and assess Kinetic and Kinematic characteristics between current design and new design of Vanguard High Flex Rotating Platform Knee Systems | Vanguard<br>High Flex<br>RP (New<br>Design) | Vanguard High<br>Flex RP (same<br>as control from<br>subgroup 2) | Historical/concurrent control | ROM, AKS,<br>Survivorship<br>and<br>Fluoroscopic<br>analysis, Gait<br>lab analysis,<br>patella clunk<br>and crepitus. |

<sup>\*</sup>Japanese sites will include equal number of Healthy Knees for ROM, Kinetic and Kinematic analysis.

<sup>\*\*</sup> Subgroup 4 will be initiated once the new design of Vanguard high flex RP is release.



The study will be conducted over a period of 12 to 15 years. Patients from subgroups 2 and 4 will be followed at immediate postop, 6 weeks, 6 months, 1 year, 3 years, 5 years, 7 years and 10 years.

#### **PATIENT SELECTION**

All subjects, regardless of sex, race, or geographic location, must fit into the scope of the Inclusion / Exclusion criteria to be eligible for the study. If required per applicable regulations, all participants must sign an Informed Consent to be enrolled into the study.

## **Inclusion Criteria**

In accordance with <u>Indications for Use</u> for Vanguard Complete Knee System and Vanguard High Flex Rotating Platform Knee System specifically:

- Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
- Correction of varus, valgus, or posttraumatic deformity.
- Correction or revision of unsuccessful osteotomy, or arthrodesis.

Patient selection factors to be considered also include:

• Need to obtain pain relief and improve function

- Ability and willingness of the patient to follow instructions, including control of weight and activity level
- · A good nutritional state of the patient, and
- The patient must have reached full skeletal maturity

#### **Exclusion Criteria**

In accordance with <u>Absolute and Relative Contraindications for use</u> for Vanguard Complete Knee System and Vanguard High Flex Rotating Platform Knee System.

Absolute contraindications include: infection, sepsis, osteomyelitis, and failure of a previous joint replacement.

#### Relative contraindications include:

- A. Uncooperative patient or patient with neurologic disorders who are incapable of following directions,
- B. Osteoporosis.
- C. Metabolic disorders which may impair bone formation,
- D. Osteomalacia.
- E. Distant foci of infections which may spread to the implant site,
- F. Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
- G. Vascular insufficiency, muscular atrophy, neuromuscular disease,
- H. Incomplete or deficient soft tissue surrounding the knee.

#### **ENDPOINTS**

| | SUBGROUP 2 | SUBGROUP 4 |
|------------|----------------------|----------------------|
| PRIMARY | Range of Motion at | Range of Motion at |
| ENDPOINTS* | 1 yr postop. | 1 yr postop. |
| | AKS at 1 year | AKS at 1 year post |
| | postop | ор |
| SECONDARY | At all follow-up | At all follow-up |
| ENDPOINTS | <u>visits:</u> | <u>visits:</u> |
| | Survivorship | Survivorship |
| | American Knee | American Knee |
| | Society Score. | Society Score. |
| | Range of Motion | Range of Motion |
| | Radiographic | Radiographic |
| | Assessment | Assessment |
| | Patient Satisfaction | Patient Satisfaction |
| | – EQ5D | – EQ5D |
| | Complications | - OKS |
| | including revisions | - FJS |
| | Patella Clunk and | Complications |
| | Crepitus | including revisions |
| | | Patella Clunk and |
| | | Crepitus |

<sup>\*</sup>For sample size calculations.

# PARTICIPANT POPULATION (SAMPLE SIZE)

Participant population is determined based on primary/secondary endpoints of each subgroup following superiority or non-inferiority methodologies. Minimum sample sizes are determined in order to prove the hypotheses.

# <u>Subgroup 2 - Primary Endpoint Range of Motion at 1 year postoperative</u> Superiority test

Null Hypothesis:  $H_0 = \mu_c$ 

Alternative Hypothesis:  $H_a$   $\mu_t = \mu_c + d$ 

 $\mu_t$ : mean of ROM in the trial group (Vanguard Complete Knee) at 1year postoperative.

 $\mu_c$ : mean of ROM in the control group (VG RP Knee) at 1 year postoperative.

a = 0.025 Significance Level (95% confidence)

 $\beta = 0.20$  80% Power

d = 5 (degrees) Clinically Relevant Difference in ROM based on literature and

engineering input.

 $\xi$  = 17.5 Estimate standard deviation of ROM at 1 year

postoperative. This value is based on results (preop and 1 year

postop) from literature<sup>1</sup>

N = 231

Consider lost to follow-up at 1 year postop, therefore the adjusted sample size is set as 250 knees per group (a total of 500 knees).

# <u>Subgroup 2 - Secondary Endpoint AKS at 1 year postoperative</u> Non-inferiority test

Null Hypothesis:  $H_0 = \mu_t = \mu_c$ 

Alternative Hypothesis:  $H_a$   $\mu_t = \mu_c + d$ 

 $\mu_t$ : mean of AKS score in the trial group (Vanguard Complete Knee) at 1 year postoperative.

 $\mu_c$ : mean of AKS score the control group (VG RP Knee) at 1 year postoperative.

<sup>&</sup>lt;sup>1</sup> Miner AL, Lingard EA, Wright EA, Sledge CB, Katz JN; Knee range of motion after total knee arthroplasty: how important is this as an outcome measure, <u>J Arthroplasty.</u> 2003 Apr;18(3):286-94.

a = 0.025 Significance Level (95% confidence)

 $\beta = 0.10$  80% Power

 $Z_{1-a/2} = 1.96$  $Z_{1-\beta} = 1.28$ 

d = 10 points Clinically Relevant Difference in Pain.

 $\xi$  = 15 Estimate standard deviation of AKS at 1 year postoperative. This value has been based on results from Biomet studies

N = 48

Consider possible lost to follow-up at 1 year postop, therefore the adjusted sample size is set as 51 knees per group. The final sample size for subgroup 2 is larger of the two sample sizes: 250 knees per group.

Therefore there will be 250 Vanguard Complete Knee will be compared to 250 Vanguard High Flex RP knee for subgroup 2 study.

Due to unknown release schedule for new designed VG High Flex RP Knee, sample size of subgroup 4 will be determined at time of the product release. Nevertheless the sample size will be determined based on the comparison to results of 250 VG High Flex RP knee of current design from subgroup 2.

## **RANDOMIZATION**

For subgroup 2 study, patients will be randomized to receive Vanguard Complete Knee (trial group), or Vanguard High Flex RP Knee (control group). Patients have an equal opportunity of being assigned to the trial group or control group. The randomization will occur via a random number generator (manual or computer). The doctor or other health care professional does not choose the participants for each group. For Patients satisfying inclusion criteria, randomization will occur by retrieving the next randomly generated group assignment.

## INSTITUTIONS

There will be a maximum of 8 sites from Korea and Japan in subgroup 2. The number of sites for subgroup 4 will be determined once new design of Vanguard High Flex RP is released.

#### PARTICIPANT DATA MANAGEMENT

The following table summarizes data collection required during the course of the study.

| SUBGROUP 2 | PRE-<br>Op | SURGERY | IMMEDIATE POST-OP | 3<br>MO | 6<br>MO | 1<br>YR | 3<br>YR | 5<br>YR | 7<br>YR | 10<br>YR |
|---|---|---|---|---|---|---|---|---|---|---|
| Informed<br>Consent | Х | | | | | | | | | |
| Demographic | Х | | | | | | | | | |

05<sup>th</sup>-Nov-2014 7

| and Historical<br>Record | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Preoperative AKS | X | | | | | | | | | |
| Operative<br>Record | | X | | | | | | | | |
| Immediate Post-Operative Radiographic Assessment (Bench Mark) | | | x | | | | | | | |
| Postoperative AKS (Including ROM) | | | | х | х | х | Х | Х | Х | x |
| Patella Clunk and Crepitus | | | | X | X | X | | | | |
| EQ5D | | | | Х | Х | X | Х | Χ | Х | Х |
| Radiographic<br>Assessment | | | | Х | X | X | x | X | X | х |
| Complications & Revisions | | | | Anytime | | | | | | |

| SUBGROUP 4 | PRE-<br>Op | SURGERY | IMMEDIATE POST-OP | 3<br>MO | 6<br>MO | 1<br>YR | 3<br>YR | 5<br>YR | 7<br>YR | 10<br>YR |
|---|---|---|---|---|---|---|---|---|---|---|
| Informed<br>Consent | X | | | | | | | | | |
| Demographic<br>and Historical<br>Record | X | | | | | | | | | |
| Preoperative<br>AKS | X | | | | | | | | | |
| Operative<br>Record | | X | | | | | | | | |
| Immediate Post-<br>Operative<br>Radiographic<br>Assessment<br>(Bench Mark) | | | x | | | | | | | |
| Postoperative<br>AKS (Including<br>ROM) | | | | x | x | X | X | X | X | x |
| Patella Clunk and Crepitus | | | | X | X | X | X | X | X | Х |
| EQ5D/SF36 | | | | X | X | Χ | Χ | Х | X | X |
| Radiographic<br>Assessment | | | | Х | Х | X | X | X | X | X |
| Complications & Revisions | | | | Anytime | | | | | | |

#### PARTICIPANT EVALUATION SCHEDULES

All study Participants are expected to return for clinical, kinetic and kinematic analysis if any and radiographic evaluation at specific follow-up intervals. The following table summarizes the schedule for post-operative follow-up time intervals:

| Evaluation Schedule | | |
|---|---|---|
| Interval | Follow-Up<br>Window | Months Post-Op Range |
| Immediate Post-<br>Op | ± 2 weeks | Immediate post-<br>op<br>< 2 weeks |
| 3 month follow-up | ± 1 month | 2-4 |
| 6 month follow-up | ± 1 month | 5-7 |
| 1 year follow-up | ± 2 months | 10-14 |
| 3 year follow-up | ± 3 months | 33-39 |
| 5 year follow-up | ± 3 months | 57-63 |
| 7 year follow-up | ± 3 months | 81-87 |
| 10 year follow-up | ± 3 months | 117 - 123 |

# **COMPLICATIONS (ADVERSE EVENTS)**

All adverse events, device related (see Risk Analysis Section) or non-device related, are to be recorded. Anticipated adverse events are defined, but not limited to, the following:

- Operative side knee manipulations or injections
- Operative side dislocations
- Operative side aspiration of joint fluids
- Falls
- Accidents- motor vehicle, motorcycle, ATV, etc.
- Death
- Any event in which the subject requires hospitalization or outpatient
  medical attention, including but not limited to: myocardial infarction,
  cerebral vascular accident, pulmonary emboli, gastrointestinal disorders,
  or a new diagnosis of a chronic condition (lung disease, renal disease,
  cancer, diabetes mellitus, hematological abnormalities, etc.).

# RADIOGRAPHIC PROTOCOL

## 1. Radiographic Views

The study requires a standard anteroposterior view, mediolateral view, and a skyline patellar view.

# 2. Reviewer

The study investigator will assess his own patient's radiographs.

# 3. Assessment Procedure

- Assessments will be recorded on the following two radiographic assessment reports:
  - Form XR100 (immediate post-operative)
  - Form XR200 (6 week, 6 month, 1 year, 3 year, 5 year, 7 year and 10 year.
- The radiographic films will be marked for measurements as described in the following "Measurement angles and reference points" section of this document. These "marked" radiographs will be used to determine the implant femoral flexion angle (α), tibial angle (β), total valgus angle (Ω), tibial angle (σ), and femoral flexion (γ).
- The immediate post-operative film will be used as an index for subsequent follow-up assessments.

The radiographic assessment definitions are as follows:

Anteroposterior Radiograph:

This radiographic view can be obtained with the participant in the standing or recumbent position.

Mediolateral Radiograph:

This radiographic view can be obtained with the participant in the standing or recumbent position.

Skyline Radiograph:

This radiograph view can be obtained with the patello-femoral joint in flexion

Radiolucency or Radiolucent Lines:

A radiographic clearing or line not exceeding 2mm in width at the bone/cement or cement/implant interface

Osteolysis:

A progressive radiolucency > 2mm in *two or more* zones not present on immediate postoperative radiographs and/or a bony destructive lesion that is progressive in nature.

• Migration/Subsidence:

A component migration of > 3 mm or > 3° as compared to immediate post-operative radiographs is considered a failure.

## **DATA COLLECTION**

All sites will be required to complete and submit case report forms on Biomet's online database, Joint Assist 2.0, in a timely manner. Forms will be monitored for completeness and accuracy.

Further, it is imperative that the investigator answers all questions on the case report forms. All data should be accurate, indelible, legible, dated on the date of entry, and signed by initials, and/or formal signature by the authorized personnel documenting the data.

#### **MONITORING PLAN**

Prior to commencing the study the Monitor will provide the investigators with the necessary information to enable him/her to carry out his responsibilities. This information includes but not limited to:

• Investigator Brochure i.e. study protocol, investigator responsibilities, device information, etc.

- Ethical Committee Approval Information.
- Case Report Forms.
- Patient Consent Forms
- EDC user manual

The monitor of the evaluation periodically reviews the post-operative follow-up dates on all subjects for each evaluator. A follow-up schedule is then sent to each investigator, which illustrates any follow-up, reports which are due or missing. Every effort is made to assure that follow-up reports are completed in a timely manner, including contacting the evaluator by post, telephone or by personal visit when necessary. Also, during the course of the evaluation, the monitor will conduct periodic discussions with the investigator or staff to ensure that the evaluation is being conducted in accordance with the protocol. The monitor will maintain records of each visit or discussion.

## **CONFIDENTIALITY**

To ensure study patients' privacy, all patients will be identified by unique identification numbers. All case report forms will only include patient IDs. It is the responsibility of the investigator to maintain a list of patient identification and Joint Assist 2.0 ID numbers.

Further the Joint Assist database is restricted, allowing a doctor to only view and enter data from his own patients. User authentication is required to view research data. The data is transmitted to a centralized database through a secured (SSL) channel on the Internet. Data in transit is in 128-bit encryption. The access to the centralized database is limited to those who are responsible for maintaining the database.

#### **RISK ANALYSIS**

This clinical study is to collect data on the Vanguard DD RP Knee, which is intended to help the participant gain mobility and decrease pain. Risks associated with this knee system include general surgical and knee arthroplasty risks. Due to the investigational nature of the system, there are unknown risks.

#### **General Surgical Risks**

As with any surgical procedure, there are risks involved with total joint replacement surgery. Potential adverse events include, but are not limited to: early or late infection perhaps necessitating device removal; component dislocation; damage to nerves and blood vessels; fracture of the bone or device; device loosening; allergic reactions to the metallic devices; phlebitis; long-term swelling; pulmonary embolization; and delayed wound healing. Other potential adverse effects include: prolonged illness; hematoma; wound dehiscence and/or drainage; the need for blood transfusions and/or further surgery; or permanent pain; deformity; and inconvenience. Risks associated with the anesthetic are those such as permanent brain damage, pneumonia, blood clots, and heart attack. Rarely some adverse events may be fatal. These possible adverse events are not unique to the Vanguard™ RP System and, as stated above, may occur with any total joint replacement surgery.

As with any joint replacement post-operative activity, limitations may be imposed

depending upon the participant's age, general health, baseline (pre-operative) activity level and baseline (pre-operative) condition of the knee and other joints.

# Potential Risks Associated with Vanguard™ RP Knee System

The safety and efficacy of the Vanguard™ RP Knee System has not been thoroughly demonstrated clinically, participants participating in the study may be subject to increased risks and/or adverse events including, but not limited to:

- 1. Material sensitivity reactions
- 2. Early or late post-operative infection and/or allergic reaction
- 3. Intra-operative bone perforation or fracture
- 4. Loosening or migration of implants
- 5. Periarticular calcification or ossification, with or without impediment of joint mobility
- 6. Inadequate range of motion
- 7. Dislocation or subluxation of device
- 8. Fatigue fracture of components
- 9. Fretting or corrosion of implant interfaces
- 10. Wear and/or deformation of articulating surfaces
- 11. Valgus/Varus deformity
- 12. Transient peroneal palsy secondary to surgical manipulation and increased joint movement
- 13. Patellar tendon rupture and ligamentous laxity
- 14. Intra-operative or post operative bone fracture
- 15. Post operative pain and/or delayed wound healing
- 16. Inadequate lubrication
- 17. Implant of the device may require a more demanding implantation procedure with greater surgical exposure and prolonged surgical time
- 18. Damage to surrounding tissues, cartilage, or tendons
- 19. Long term swelling
- 20. Excessive bleeding
- 21. Instability

## Minimization of Risk

With the increased understanding of failure modes for mobile bearing knees, preclinical testing and clinical results found in the literature, it is believed that none of the previously mentioned adverse events will occur in significant numbers. This investigational plan has reduced the potential risk to the participant through the following methods:

- By defining a participant population that limits the exposure of the device to participants conforming to the proposed indications, exclusions, and age requirements
- 2. The surgical technique has been developed to help eliminate potential operative difficulties.

#### **REFERENCES**

- 1. Mulholland, S.J. and U.P. Wyss, *Activities of daily living in non-Western cultures:* range of motion requirements for hip and knee joint implants. Int J Rehabil Res, 2001. **24**(3): p. 191-8.
- 2. Thambyah, A., J.C. Goh, and S.D. De, *Contact stresses in the knee joint in deep flexion*. Med Eng Phys, 2005. **27**(4): p. 329-35.
- 3. Masashi Tamaki, Tetsuya Tomita, Takaharu Yamazaki, William J. Hozack, Hideki Yoshikawa, and Kazuomi Sugamoto, *In Vivo Kinematic Analysis of a High-Flexion Posterior Stabilized Fixed-Bearing Knee Prosthesis in Deep Knee-Bending Motion;* The Journal of Arthroplasty Vol. 23 No. 6 2008
- 4. Kouichi Kanekasu, Scott A. Banks, Shigeru Honjo, Osanari Nakata, and Hiromi Kato; Fluoroscopic Analysis of Knee Arthroplasty Kinematics During Deep Flexion Kneeling; The Journal of Arthroplasty Vol. 19 No. 8 2004

Alberto A. Bolanos, Wayne A. Colizza, Peter D. McCann, Robert S. Gotlin, Mary E. Wootten, Barbara A. Kahn, and John N. Insall, *A Comparison of Isokinetic Strength Testing and Gait Analysis in Patients With Posterior Cruciate-Retaining and Substituting Knee Arthroplasties*; The Journal of Arthroplasty Vol. 13 No. 8 1998